CLINICAL TRIAL: NCT05110014
Title: Substudy of Protocol NCT03843957: Effect of mPATH on Screening for Depression, Fall Risk, and Safety
Brief Title: Substudy of Protocol NCT03843957 - Effect of mPATH on Screening for Depression, Fall Risk, and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00048919.sub; R01CA218416 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-02

CONDITIONS: Depression
Keywords: Fall risk; Intimate partner violence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Care Office Visits (Other): The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Interventions: Other: Primary Care Office Visits

INTERVENTIONS:
Other: Primary Care Office Visits — mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence

SUMMARY:
This is a sub-study for data analysis of data collected as part of the larger randomized controlled trial "Effectiveness and Implementation of mPATH-CRC" (NCT03843957) to determine if self-administered screening with an iPad increases the detection of patients with depression, falls, and intimate partner violence.

DETAILED DESCRIPTION:
As part of the parent study (NCT0343957), investigators developed an iPad program called mPATH that patients use at their primary care clinician's office to encourage colorectal cancer screening. To encourage practices to use mPATH with every patient, the investigators included in the program the health system's required screening items for depression, fall risk, and intimate partner violence, thereby offloading this routine task from clinical staff. It is possible that mPATH will increase detection of depression, fall risk, and intimate partner violence because: 1) mPATH systematically asks these screening items of all patients, and 2) patients may feel more comfortable answering these items on an iPad survey than during an in-person interview.

To determine the effect of mPATH on the performance of this screening, investigators will examine a limited use dataset comparing the 2 months before a clinic started using mPATH to the 2 months after the clinic began using mPATH. Because clinics may need some time to fully adopt mPATH, investigators will exclude the first two weeks following the launch of mPATH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Completed a provider visit at the study clinic during the 60 days prior to the clinic launching the mPATH program (the "pre" time period), or completed a provider visit at the study clinic during days 14 - 73 after the launch of mPATH (the "post" time period)
* Have a preferred language of English or Spanish

Exclusion Criteria:

• Requiring a language interpreter for a language other than Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23026 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, MS, Principal Investigator — Wake Forest Baptist Health Sciences
Locations (1):
- Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Before mPATH Launch: The number of participants screened prior to the mPATH intervention.
  The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Primary Care Office Visits: mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence
- After mPATH Launch: The number of participants screened after MPATH intervention.
  The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Primary Care Office Visits: mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence
Period: Overall Study
Arm/Group | Before mPATH Launch | After mPATH Launch
Started | 12239 | 10787
Completed | 12239 | 10787
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Primary Care Office Visits - Before mPATH; Primary Care Office Visits - After mPATH: The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Primary Care Office Visits: mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence
- Total: Total of all reporting groups
Arm/Group | Primary Care Office Visits - Before mPATH | Primary Care Office Visits - After mPATH | Total
Number analyzed (Participants) | 12239 | 10787 | 23026
Age, Continuous [Mean (Full Range); unit: years] | 60.2 [18 to 102] | 59.0 [18 to 102] | 59.7 [18 to 102]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7030 | 6312 | 13342
  Male | 5209 | 4475 | 9684
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 387 | 357 | 744
  Not Hispanic or Latino | 11677 | 10287 | 21964
  Unknown or Not Reported | 175 | 143 | 318
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 161 | 163 | 324
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1640 | 1458 | 3098
  White | 9876 | 8666 | 18542
  More than one race | 175 | 143 | 318
  Unknown or Not Reported | 387 | 357 | 744
Region of Enrollment [Number; unit: participants]
  United States | 12239 | 10787 | 23026
Primary Health Insurance [Count of Participants; unit: Participants]
  Commercial | 5382 | 4962 | 10344
  Medicaid | 401 | 377 | 778
  Medicare | 5705 | 4817 | 10522
  Uninsured | 462 | 367 | 829
  Other | 289 | 264 | 553
Primary Care Practices [Count of Participants; unit: Participants]
  Practice A | 1935 | 1730 | 3665
  Practice B | 1574 | 1868 | 3442
  Practice C | 1943 | 1877 | 3820
  Practice D | 2866 | 1873 | 4739
  Practice E | 2215 | 2170 | 4385
  Practice F | 1706 | 1269 | 2975

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Screening Positive for Depression, Fall Risk or Intimate Partner Violence - Pre mPATH Use
Description: The primary outcome will be the proportion of patients seen in each time period ("pre" vs. "post") who screen positive for depression, fall risk, or intimate partner violence. The "pre" time period will be Days -60 to -1 (the 60 day period before mPATH Launch). Screening positive for depression will be a score of 3 or greater on the Patient Health Questionnaire-2. Screening positive for fall risk will be answering "yes" to having a device to assist with mobility and/or having fallen in the last year. Screening positive for intimate partner violence will be answering yes to any of the health system's three questions about safety in the home.
Time Frame: 2 months prior to use of intervention
Population: Investigators prefer not to identify the practices by types: 1) Investigators do not hypothesize there will be any difference in effect by practice type and naming the clinics by type could make a reader assume investigators were looking for a 'practice-type' effect), and 2) not identifying which practices further protects the confidentiality of the practices. Overall number = 1,067 is the overall number of participants that were positive out of the 12,239 before mPATH intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Care Practices: The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Primary Care Office Visits: mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 12239
Participants
  Practice A: number analyzed (Participants) | 1067
  Practice A | 224
  Practice B: number analyzed (Participants) | 1,067
  Practice B | 94
  Practice C: number analyzed (Participants) | 1,067
  Practice C | 55
  Practice D: number analyzed (Participants) | 1,067
  Practice D | 165
  Practice E: number analyzed (Participants) | 1,067
  Practice E | 265
  Practice F: number analyzed (Participants) | 1,067
  Practice F | 264

2. Primary Outcome: Number of Participants Screening Positive for Depression, Fall Risk or Intimate Partner Violence - Post mPATH Use
Description: The primary outcome will be the proportion of patients seen in each time period ("pre" vs. "post") who screen positive for depression, fall risk, or intimate partner violence. The "post" time period will be days 14 to 73 (the 60 day period commencing 2 weeks after mPATH Launch). Screening positive for depression will be a score of 3 or greater on the Patient Health Questionnaire-2. Screening positive for fall risk will be answering "yes" to having a device to assist with mobility and/or having fallen in the last year. Screening positive for intimate partner violence will be answering yes to any of the health system's three questions about safety in the home.
Time Frame: 2 months after use of intervention
Population: Positive screenings for composite outcomes (depression, fall risk, intimate partner violence) were reported in individual medical practices - 3 family medicine and 3 internal medicine practices. The count of participants = 2,102 is the overall number of participants that were positive out of the 10,787 after mPATH intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Care Office Visits: The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Primary Care Office Visits: mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence
Arm/Group | Primary Care Office Visits
Number analyzed (Participants) | 10787
Participants
  Practice A: number analyzed (Participants) | 2102
  Practice A | 509
  Practice B: number analyzed (Participants) | 2102
  Practice B | 463
  Practice C: number analyzed (Participants) | 2102
  Practice C | 235
  Practice D: number analyzed (Participants) | 2102
  Practice D | 242
  Practice E: number analyzed (Participants) | 2102
  Practice E | 418
  Practice F: number analyzed (Participants) | 2102
  Practice F | 235

3. Secondary Outcome: Number of Participants Screening Positive for Depression Using Patient Health Questionnaires (PHQ-2 Score of 3 or Greater)
Description: The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past two weeks. Screen positive for depression using the PHQ-2 items. PHQ-2 score obtained by adding score for each question (total points). A PHQ-2 score ranges from 0-6. If the score is 3 or greater, major depressive disorder is likely.
Time Frame: 2 months before and 2 months after using intervention
Population: The number includes the actual number of participants that were analyzed (2 months before and 2 months after the intervention) out of the total of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Office Visits
Number analyzed (Participants) | 23026
Participants
  Before intervention: number analyzed (Participants) | 12239
  Before intervention | 188
  After intervention: number analyzed (Participants) | 10787
  After intervention | 450

4. Secondary Outcome: Number of Participants Screening Positive for Moderately Severe or Severe Depression Using Patient Health Questionnaires (PHQ-9 Score Greater Than 14)
Description: The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ-9 score obtained by adding score for each question (total points). Total scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: 2 months before and 2 months after using intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Office Visits
Number analyzed (Participants) | 23026
Participants
  Before Intervention: number analyzed (Participants) | 12239
  Before Intervention | 82
  After intervention: number analyzed (Participants) | 10787
  After intervention | 206

5. Secondary Outcome: Number of Participants Screening Positive for Severe Depression Using Patient Health Questionnaires (PHQ-9 Score Greater Than 19)
Description: as for outcome 4
Time Frame: 2 months before and 2 months after using intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Office Visits
Number analyzed (Participants) | 23026
Participants
  Before intervention: number analyzed (Participants) | 12239
  Before intervention | 28
  After intervention: number analyzed (Participants) | 10787
  After intervention | 86

6. Secondary Outcome: Number of Participants With a Patient Health Questionnaires (PHQ-9 Score Greater Than 14) and Not Currently Taking a Medication for Depression.
Description: as for outcome 4
Time Frame: 2 months before and 2 months after using intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Office Visits
Number analyzed (Participants) | 23026
Participants
  Before Intervention: number analyzed (Participants) | 12239
  Before Intervention | 63
  After intervention: number analyzed (Participants) | 10787
  After intervention | 139

7. Secondary Outcome: Number of Participants Who Report Thoughts of Self Harm - Patient Health Questionnaire (PHQ-9) in All Practices
Description: This is measured by the screening question on suicide risk on the PHQ-9: "Thoughts that you would be better off dead or of hurting yourself in some way."
Time Frame: 2 months before and 2 months after using intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Primary Care Office Visits (Pre Intervention); Primary Care Office Visits (Post Intervention): The limited use dataset will contain the following data elements for each completed patient visit:
  * Date of clinic visit (where each date is indicated by a number relative to the clinic's Launch Date)
  * Clinic (designated by a unique study clinic identifier)
  * Type of visit completed (for example, new patient visit, return patient visit, annual exam)
  * Patient age
  * Patient gender
  * Patient race/ethnicity
  * Patient primary insurance
  * Nursing staff who roomed the patient (designated by a unique study identifier)
  * Whether patient used mPATH-CheckIn program (Y/N)
  * Whether nursing staff used mPATH Nursing Module to transmit mPATH data to electronic health record (Y/N)
  * Whether patient has a diagnosis of depression in the problem list in the EHR (Y/N)
  * Whether patient has an antidepressant medication listed in the active medication list ( (Y/N)
  * Results of depression screening items
  * Results of fall risk screening items
  * Results of safety at home screening items
  Primary Care Office Visits: mPATH iPad program that contains self-administered screening items for depression, fall risk, and intimate partner violence
Arm/Group | Primary Care Office Visits (Pre Intervention) | Primary Care Office Visits (Post Intervention)
Number analyzed (Participants) | 1067 | 2102
Participants | 39 | 116

8. Secondary Outcome: Number of Participants Screening Positive for Fall Risk at Home in All Practices
Description: Screen positive for fall risk at home. In addition, the outcomes below will be assessed:
  * Have fallen in last 6 months
  * Have had a fall with injury
Time Frame: 2 months before and 2 months after using intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Office Visits (Pre Intervention) | Primary Care Office Visits (Post Intervention)
Number analyzed (Participants) | 1067 | 2102
Participants | 907 | 1692

9. Secondary Outcome: Number of Participants Screening Positive for Intimate Partner Violence in All Practices
Description: Screen positive for safety concerns at home. In addition, the outcome below will be assessed:
  * Report that conflicts turn into fights
Time Frame: 2 months before and 2 months after using intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Office Visits (Pre Intervention) | Primary Care Office Visits (Post Intervention)
Number analyzed (Participants) | 1067 | 2102
Participants | 10 | 310

ADVERSE EVENTS:
Description: Adverse events were not collected for this portion of the study
Arm/Group | Primary Care Office Visits (Pre Intervention) | Primary Care Office Visits (Post Intervention)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT05110014/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT05110014/ICF_001.pdf